CLINICAL TRIAL: NCT02401776
Title: An Evaluation of the Heart Rate, Blood Pressure and Repolarization Effects of an Energy Drink as Compared to Coffee
Brief Title: Effect of Caffeine on Heart Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Robert M. Brothers, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2014-03-0069
Record Dates: First submitted 2014-05-20; First posted 2015-03-30 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Fatigue; Tachycardia
Keywords: heart rate; blood pressure; caffeine; energy drink
MeSH Terms: conditions — Fatigue; Tachycardia | interventions — Coffee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- small dose monster energy drink (Experimental): This will be a small dose of monster energy drink
  Interventions: Dietary Supplement: Monster Energy Drink; Dietary Supplement: Coffee
- medium dose monster energy drink (Experimental): This will be a medium dose of monster energy drink
  Interventions: Dietary Supplement: Monster Energy Drink; Dietary Supplement: Coffee
- coffee (Active Comparator): This will be a coffee group and will drink Starbuck's K-cup Breakfast Blend. This will be mixed according to packing instructions and will be given at a dose of 2mg caffeine/kg body weight (equivalent to approximately one 11 ounce cup of coffee for a person weighing 75 kg).
  Interventions: Dietary Supplement: Monster Energy Drink; Dietary Supplement: Coffee

INTERVENTIONS:
Dietary Supplement: Monster Energy Drink — Small Dose of Monster energy drink. This will be given at a dose of 2mg caffeine/kg body weight (equivalent to approximately one 16 ounce can of monster energy drink for a person weighing 75 kg).
Dietary Supplement: Monster energy drink — Medium Dose of Monster Energy Drink. This will be given at a dose of 3 mg caffeine/kg body weight (equivalent to approximately one 24 ounce can of monster energy drink for a person weighing 75 kg).
Dietary Supplement: Monster Energy Drink — Monster energy drink. This will be given at a dose of 3mg caffeine/kg body weight (equivalent to approximately one 24 ounce can of monster energy drink for a person weighing 75 kg).
Dietary Supplement: Coffee — Coffee. This will be given at a dose of 2mg caffeine/kg body weight (equivalent to approximately one 8 ounce cup of coffee drink for a person weighing 75 kg).

SUMMARY:
* The primary objective of this study is to assess the effect of an energy drink on ventricular repolarization as measured by the interval between the cardiac Q wave and the cardiac T wave (QT interval)obtained from the body surface ECG.
* The secondary objective is to assess the effects of an energy drink on heart rate and blood pressure (hemodynamic effects).

To place the observed changes in context, comparison will be made to a commonly consumed drink, coffee: Starbuck's K-cup Breakfast Blend.

DETAILED DESCRIPTION:
This study will assess cardiac repolarization before and after three conditions each of which will involve the subject drinking beverages of varying caffeine content.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI between 24 - 29

Exclusion Criteria:

* Resting heart rate below 60 bpm
* Resting heart rate above 88 bpm
* Cardiovascular or metabolic disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
QT interval will be measured in msec | 19 hrs
  The investigators will be measuring cardiac QT interval before (baseline) and for 5 hours post beverage consumption. The measurements will be made in msec.

SECONDARY OUTCOMES:
Heart rate will be measured as beats per minute. | 19 hrs
  The investigators will be measuring cardiac heart rate before (baseline) and for 5 hours post beverage consumption. The measurements will be made as beats per minute.
Blood Pressure will be measured in the brachial artery as mmHG | 19 hrs
  The investigators will be measuring artery blood pressure before (baseline) and for 5 hours post beverage consumption. The measurements will be made as mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Brothers, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- Environmental and Autonomic Physiology Laboratory; University of Texas at Austin, Austin, Texas, United States